CLINICAL TRIAL: NCT06155409
Title: Safety and Performance of the SpineVision Hexanium ACIF in the Treatment of Cervical Spine Degenerative Disc Disease in Skeletally Mature Patients - HEXANIUM ACIF Study
Brief Title: Safety and Performance of the SPINEVISION Hexanium ACIF in the Treatment of Cervical Spine Degenerative Disc Disease
Status: Active, not recruiting | Type: Observational
Sponsor: SPINEVISION SAS (Industry)
Collaborators: EVAMED (Other)
Responsible Party: Sponsor
Other Study IDs: SV004
Record Dates: First submitted 2023-11-23; First posted 2023-12-04 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Intervertebral Disc Degeneration
Keywords: Spine; Arthrodesis; Stabilization; Neck Disability Index; Visual Analogue Score; Cervical; Fusion
MeSH Terms: conditions — Intervertebral Disc Degeneration; Ankylosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Anterior cervical interbody fusion — Anterior cervical interbody fusion indicates a surgical approach in the cervical spine to fuse the discal space between two vertebrae. These are joined by removing the disc and placing a cage in its place to restore the vertebral height.

SUMMARY:
The goal of this observational study is to confirm the safety and efficacy of the Hexanium ACIF system in the treatment of skeletally mature patients suffering from degenerative disc disease (disease that occurs when the spinal disk breaks down) at the cervical spine level (C3-C7).

Part of their standard of care, participants will be questioned on their neck and arm pains, their disability and if they have encountered any adverse effects since the Hexanium ACIF system implant surgery. Those data will be collected up to twenty four (24) months after the Hexanium ACIF system implant surgery.

DETAILED DESCRIPTION:
The Hexanium ACIF study is a multicentric, non-randomized, ambispective, post market clinical follow-up study. This means that either subjects already implanted with the Hexanium ACIF system (retrospective subjects) or subjects planned for treatment with the Hexanium ACIF system (prospective subjects) can be enrolled in hte study.

Standard of care subjects data up to twenty four (24) months post Hexanium ACIF system implant procedure will be collected; key data include neck and arm Visual Analogue Score (VAS), Neck Disability Index (NDI) score, and adverse events.

Data will be collected at Month 2, Month 6, Month 12 and Month 24 post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient planned for Hexanium ACIF system implant or patient implanted with Hexanium ACIF system (not prior July 2020)
* Patient of 18 years old or more
* Patient has provided signed informed consent, or did not oppose to his/her data collection, per local regulation

Exclusion Criteria: contra-indication

* Infection, local to the operative site
* Signs of local inflammation
* Fever or leukocytosis
* Morbid obesity
* Pregnancy
* Paediatric cases, or patient still having general skeletal growth
* Spondylolisthesis unable to be reduced to Grade I
* Suspected or documented allergy or intolerance to metal
* Any case where the implant components selected for use would be too large or too small to achieve a successful result
* Any patient having inadequate tissue coverage over the operative site or inadequate bone stock or quality
* Any patient in which implant utilization would interfere with anatomical structures or expected physiological performance
* Prior fusion at the level to be treated
* Any case not needing a bone graft or fusion
* Any abnormality present which affects the normal process of bone remodelling including, but not limited to severe osteoporosis involving spine, bone absorption, osteopenia, primary or metastasis tumours involving the spine, active infection at the site or certain metabolic disorders affecting osteogenesis
* Any other condition which would preclude the potential benefit of spinal implant surgery, such as the presence of tumours or congenital abnormalities, fracture local to operating site, elevation of segmentation rate unexplained by other diseases, elevation of white blood count (WBC), or marked left shift in the WBC differential count
* Mental illness
* Any patient unwilling to cooperate with postoperative instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients elligible for treatment or already treated with the Hexanium ACIF system device will be offered to participate in the study; this applies to primary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of serious adverse device and/or procedure related events | Month 24
  Rate of serious adverse events related to the study device and / or surgical implant procedure will be analyzed and compared to the state of the art.
Change of the Neck Disability Index (NDI) | Month 12
  Neck Disability Index (NDI) mean score at Month 12 will be compared to Neck Disability Index (NDI) mean score at baseline.
  Neck Disability Index (NDI) score varies between 0% and 100%, with highest score as worst outcome.

SECONDARY OUTCOMES:
Fusion success | Month 2, month 6, month 12 and month 24
  Fusion rate will be analyzed and compared to the sate of the art.
Change of the Neck Disability index (NDI) | Month 2, month 6, month 12 and month 24
  Mean Neck Disability Index (NDI) score evolution will be analyzed. Neck Disability Index (NDI) score varies between 0% and 100%, with highest score as worst outcome.
Change of the neck and arm Visual Analogue Score (VAS) | Month 2, month 6, month 12 and month 24
  Neck and arm Visual Analogue Score (VAS) assessments will be analyzed. Visual Analogue Score (VAS) is a pain scoring, with score varying from 0 (no pain) to 10 (worst pain, unbearable, excrutiating pain)
Incidence of revision surgery at implant site | Month 2, month 6, month 12 and month 24
  Rate of revision surgery at implant site will be analyzed and compared to the state of the art.

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Lucas, Doctor, Principal Investigator — Centre Hospitalier de l'Europe
Locations (6):
- France (6):
  - Clinique du Dos Terrefort, Bordeaux
  - Centre Hospitalier Privé de l'Europe, Le Port-Marly
  - CHRU de Nancy, Nancy
  - Polyclinique Majorelle, Nancy
  - Hôpital Privé du Dos Francheville, Périgueux
  - Hôpital Robert Schuman - UNEOS, Vantoux

IPD SHARING:
Plan to Share IPD: No